CLINICAL TRIAL: NCT00109161
Title: A Phase II Randomized, Double-Blinded, Placebo-Controlled, Multi-Center Study of Subcutaneous Daclizumab in Patients With Active, Relapsing Forms of Multiple Sclerosis
Brief Title: Study of Subcutaneous Daclizumab in Patients With Active, Relapsing Forms of Multiple Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PDL BioPharma, Inc. (Industry)
Organization: Facet Biotech (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DAC-1012
Record Dates: First submitted 2005-04-22; First posted 2005-04-25 (Estimated); Last update posted 2008-08-05 (Estimated); Status verified 2008-08

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis, MS, CNS, Daclizumab
MeSH Terms: conditions — Multiple Sclerosis | interventions — Daclizumab

INTERVENTIONS:
Drug: Daclizumab (Anti-CD25 Humanized Monoclonal Antibody)

SUMMARY:
This research study is being conducted in the U.S. and Europe to evaluate the safety and efficacy of daclizumab for the treatment of multiple sclerosis (MS).

DETAILED DESCRIPTION:
PDL BioPharma, Inc. was formerly known as Protein Design Labs, Inc.

ELIGIBILITY:
Inclusion Criteria:

* Male or female age 18 to 55 years, inclusive.
* Diagnosis of MS by McDonald criteria.
* EDSS <7.0.
* On stable IFN-beta regimen for at least 6 months.
* The occurrence of either of the following within 9 months prior to screening: ≥1 MS relapse OR A qualifying MRI, defined as an MRI that showed at least one confirmed Gd-CEL of the brain or spinal cord, was performed independently of the study while the patient was on a stable IFN-beta regimen, and is deemed acceptable by the central reader.
* For females, women of non-childbearing potential or women of childbearing potential who provide a negative serum pregnancy test at screen and within 24 hours of first dose of study drug, and who agree to use effective contraception during the Treatment and Follow-up periods of the study.
* Willing and able to comply with the protocol, provision of informed consent in accordance with institutional and regulatory guidelines, and, for US sites only, authorization to use protected health information.

Exclusion Criteria:

* Pregnant or breast-feeding woman.
* Non-ambulatory patient.
* Clinically significant abnormality on screening ECG.
* Malignancy within the past 5 years, except for adequately treated non-melanoma skin carcinoma or in situ carcinoma of the cervix.
* History of HIV infection, positive serology for HBV (hepatitis B virus) or HCV (hepatitis C virus).
* Varicella (VZV) or herpes zoster virus infection, or any severe viral infection, within 6 weeks before screening or exposure to VZV within 21 days of screening.
* Abnormal hematology, as defined by the following laboratory values: *Hemoglobin ≤8.5 g/dL, *Lymphocytes ≤1.0 x 10^9/L, *Platelets ≤100 x 10^9/L, *Neutrophils ≤1.5 x 10^9/L.
* Significant organ dysfunction, including but not limited to cardiac, renal, liver, non-MS related CNS, pulmonary, vascular, gastrointestinal, endocrine, or metabolic dysfunction, or other disease or condition, which in the opinion of the PI (principal investigator) would make the patient an unsuitable candidate for the study. Guidelines for levels of unacceptable dysfunction include: *creatinine ≥1.6 mg/dL; *AST and ALT ≥2.5 times upper limit of normal (ULN); *alkaline phosphatase ≥2.5 times ULN; *history of myocardial infarction, congestive heart failure, or arrhythmias within 6 months prior to randomization.
* Use of any of the following: *Any of the following types of live virus vaccine from 4 weeks before randomization: measles/mumps/rubella vaccine, varicella zoster virus vaccine, oral polio vaccine, and nasal influenza vaccine. Use of these vaccines, however, by household contacts does not affect the eligibility of patients to enroll or continue in the study; *Systemic corticosteroids, adrenocorticotropic hormone, or plasma exchange within 4 weeks before the baseline MRI scan (no more than 72 hours before Day 0); *Azathioprine, mycophenolate mofetil, methotrexate, glatiramer acetate, or intravenous immune globulin within 6 months before randomization; *An immunomodulatory agent within 6 months before randomization, except for interferon-beta products required per protocol; *An investigational agent within 6 months before randomization unless this agent is non-immunomodulatory and the medical monitor or steering committee rules that its use is acceptable on the theoretical basis of a lapse of at least 5 serum half-lives since administration of the last possible dose; *A monoclonal antibody (eg, Rituxan®/ Rituximab) within 6 months before randomization; *Daclizumab at any time prior to randomization; *Cladribine, mitoxantrone, cyclophosphamide, CamPath® (alemtuzumab), natalizumab (TYSABRI®/Antegren) or other drugs targeting alpha 4 integrin, total lymphoid irradiation, or bone marrow transplant at any time
* Patients for whom MRI is contraindicated, ie, have pacemakers or other contraindicated implanted metal devices, are allergic to gadolinium, or have claustrophobia that cannot be medically managed.
* Primary progressive MS.
* Clinically unstable for 30 days before randomization (Patients who experienced a relapse, with or without steroid treatment, during the screening period may be re-screened after 30 days.)
* Elective surgery performed from 2 weeks prior to randomization or scheduled through Week 44
* Infection (viral, fungal, bacterial) requiring hospitalization or IV antibiotics within 8 weeks before randomization.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 270
Dates: Start 2005-04; Study Completion 2006-10

PRIMARY OUTCOMES:
Number of new or enlarged gadolinium contrast enhancing lesions (Gd-CELs) on monthly brain MRIs collected between Weeks 8 to 24 in daclizumab- vs. placebo-treated patients

SECONDARY OUTCOMES:
Pharmacokinetics
Immunogenicity
Clinical improvement

CONTACTS AND LOCATIONS:
Overall Officials: Richard Dickson, M.D., Principal Investigator — Wenatchee Valley Medical Center; Steven Pugh, M.D., Principal Investigator — Rockwood Clinic, PS; Daniel Wynn, M.D., Principal Investigator — Consultants in Neurology; Theodore J. Phillips, M.D., Principal Investigator — The MS Center at Texas Neurology; Joanna Cooper, Principal Investigator — Sutter East Bay Medical Foundation; James R. Storey, Principal Investigator — Upstate Clinical Research; Malcolm Gottesman, M.D., Principal Investigator — Winthrop University Hospital; Herman Sullivan, M.D., Principal Investigator — Michigan Medical P.C. Neurology; Timothy Vollmer, M.D., Principal Investigator — St. Joseph's Hospital and Medical Center, Phoenix; Jeffery Dunn, M.D., Principal Investigator — MS Hub Medical Group; S. Mitchell Freedman, M.D., Principal Investigator — Raleigh Neurology Associates; Joseph Herbert, M.D., Principal Investigator — Hospital for Joint Diseases, MS Care Center; Omar Khan, M.D., Principal Investigator — Wayne State University MS Center; Marcelo Kremenchutzky, M.D., Principal Investigator — London Health Sciences Centre; Sharon Lynch, M.D., Principal Investigator — CLMC Neurology; Alireza Minagar, M.D., Principal Investigator — Louisiana State University Health Sciences Center; Jeffrey English, M.D., Principal Investigator — The Multiple Sclerosis Center of Atlanta; Andrew Goodman, M.D., Principal Investigator — University of Rochester; Michael Kaufman, M.D., Principal Investigator — MS Center/CMC; Florian P. Thomas, M.D., Principal Investigator — St. Louis University Hospital; Clyde Markowitz, M.D., Principal Investigator — University of Pennsylvania; Jayne Martin, M.D., Principal Investigator — Michigan State University; Maria Melanson, M.D., Principal Investigator — Health Sciences Center; MaryAnn Picone, M.D., Principal Investigator — Gimble MS Center; Christopher Bever, M.D, Principal Investigator — Maryland Center for MS; Gregg G. Blevins, M.D., Principal Investigator — University of Alberta; Kasper Lloyd, M.D., Principal Investigator — MS Center at Dartmouth; Yves Lapierrre, M.D., Principal Investigator — Montreal Neurological Institute; John W. Rose, M.D., Principal Investigator — University of Utah CAMT; Michael Yeung, M.D., Principal Investigator — Foothills Medical Centre; Neil Lava, M.D., Principal Investigator — Albany Medical College; Jonathan L. Carter, M.D., Principal Investigator — Mayo Clinic; Francois Jacques, M.D., Principal Investigator — Clinique SEP/NM; William Honeycutt, M.D., Principal Investigator — Neurology Associates, P.A.; Istvan Pirko, M.D., Principal Investigator — University of Cincinnati; Ed Fox, M.D., Principal Investigator — Central Texas Neurology
Locations (36):
- United States (30):
  - St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Mayo Clinic, Scottsdale, Arizona
  - Sutter East Bay Medical Foundation, Berkeley, California
  - Neurology Associates, P.A., Maitland, Florida
  - The Multiple Sclerosis Center of Atlanta, Atlanta, Georgia
  - Consultants in Neurology, Northbrook, Illinois
  - KUMC Neurology, Kansas City, Kansas
  - Louisiana State University Health Sciences Center, Shreveport, Louisiana
  - Maryland Center for MS, Baltimore, Maryland
  - Wayne State University MS Center, Detroit, Michigan
  - Michigan State University, East Lansing, Michigan
  - Michigan Medical P.C. Neurology, Grand Rapids, Michigan
  - St. Louis University Hospital, St Louis, Missouri
  - MS Center at Dartmouth, Lebanon, New Hampshire
  - Gimble MS Center, Teaneck, New Jersey
  - Upstate Clinical Research, Albany, New York
  - Albany Medical Center, Albany, New York
  - Winthrop University Hospital, Mineola, New York
  - Hospital for Joint Diseases, MS Care Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - MS Center/CMC Meyers Park, Charlotte, North Carolina
  - Raleigh Neurology Associates, Raleigh, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - The MS Center at Texas Neurology, Dallas, Texas
  - Central Texas Neurology, Round Rock, Texas
  - University of Utah CAMT, Salt Lake City, Utah
  - MS Hub Medical Group, Seattle, Washington
  - Rockwood Clinic, PS, Spokane, Washington
  - Wenatchee Valley Medical Center, Wenatchee, Washington
- Canada (6):
  - Foothills Medical Centre-MS Research Program, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
  - Health Sciences Center, Winnipeg, Manitoba
  - London Health Sciences Centre, London, Ontario
  - Clinique SEP/NM, Gatineau, Quebec
  - Montreal Neurological Institute, Montreal, Quebec

REFERENCES:
- [Derived] Wynn D, Kaufman M, Montalban X, Vollmer T, Simon J, Elkins J, O'Neill G, Neyer L, Sheridan J, Wang C, Fong A, Rose JW; CHOICE investigators. Daclizumab in active relapsing multiple sclerosis (CHOICE study): a phase 2, randomised, double-blind, placebo-controlled, add-on trial with interferon beta. Lancet Neurol. 2010 Apr;9(4):381-90. doi: 10.1016/S1474-4422(10)70033-8. Epub 2010 Feb 15. PMID 20163990